CLINICAL TRIAL: NCT05368753
Title: Evaluation of Plasma Concentrations of Intravenous Lidocaine and Epidural Ropivacaine When Used in Combination in Major Abdominal Surgery
Acronym: LARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2021_843_0197
Record Dates: First submitted 2022-03-14; First posted 2022-05-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Abdominal Surgery by Laparotomy; Thoracic Epidural Analgesia; Analgesia; Lidocaine Adverse Reaction
Keywords: Abdominal surgery by laparotomy; thoracic epidural analgesia; Analgesia; Lidocaine Adverse Reaction
MeSH Terms: conditions — Agnosia | interventions — Blood Specimen Collection; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thoracic epidural analgesia (Experimental): Lidocaine will be injected during the anaesthetic induction and infused until the surgical closure (30 minutes before the end), then ropivacaine will be injected in the TEA at the same time and infused during 24h. The occurrence of adverse events will be monitor by a physical examination and blood samples of lidocainemia and ropivacainemia in the perioperative period
  Interventions: Other: Blood sample; Drug: Lidocain; Drug: ropivacaine

INTERVENTIONS:
Other: Blood sample — Lidocaine blood sample 30 min before the end of the surgery Lidocaine blood sample at the end of the infusion lidocaine and ropivacaine blood sample 2 h after the ropivacaine infusion of the TEA Ropivacaine blood sample 24h after the infusion of the TEA
Drug: Lidocain — Lidocaine will be injected during the anaesthetic induction and infused until the surgical closure (30 minutes before the end) The occurrence of adverse events will be monitor by a physical examination and blood samples of lidocainemia and ropivacainemia in the perioperative period.
Drug: ropivacaine — Lidocaine will be injected during the anaesthetic induction and infused until the surgical closure (30 minutes before the end), then ropivacaine will be injected in the TEA at the same time and infused during 24h. The occurrence of adverse events will be monitor by a physical examination and blood samples of lidocainemia and ropivacainemia in the perioperative period.

SUMMARY:
Thoracic epidural analgesia (TEA) is the gold standard analgesia of the laparotomy in major abdominal surgery and can be associated with intravenous lidocaine or subtituted by intravenous lidocaine when TEA is contraindicated and in order to reduce the use of the morphinics in the perioperative period.

Side effects can be paralytic ileus or nausea and vomiting and delay the enhanced recovery after surgery.

Intravenous lidocaine and TEA share several properties like anti hyperalgesia, anti inflammatory effect, intestinal process, anti tumoral effect… which suggests an additive effect of their combination that was not studied yet.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal surgery by laparotomy

Exclusion Criteria:

* laparoscopic abdominal surgery,
* TEA contraindication,
* ropivacaine contraindication
* intravenous lidocaine contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Blood lidocaine concentration (micrograms/ml) | 30 minutes before the end of surgery
  Lidocaine blood sample will be performed 30 min before the end of the surgery
blood lidocaine concentration (micrograms/ml) | at the end of the surgery (assessed up to 2 hours)
  lidocaine blood sample will be performed at the end of the infusion,
blood lidocaine and ropivacaine concentration (micrograms/ml) | at 2 hours
  lidocaine and ropivacaine blood sample 2 h after the ropivacaine infusion of the TEA,
blood ropivacaine concentration (micrograms/ml) | at 24 hours
  ropivacaine blood sample 24h after the infusion of the TEA

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No